CLINICAL TRIAL: NCT03814369
Title: Use of AmplifEYE-assisted Colonoscopy Compared to Standard Colonoscopy in Polyp and Adenoma Detection
Brief Title: AmplifEYE Colonoscopy vs Standard Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Collaborators: Our Lady of Maryknoll Hospital (Other)
Responsible Party: Principal Investigator, Sze Shun Fung, Associate Consultant, Queen Elizabeth Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: amplifeye
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Colon Polyp; Adenoma Colon; Serrated Polyp; Colonic Neoplasms
Keywords: colonoscopy; adenoma detection rate; colorectal cancer screening; new technology
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AmplifEYE colonoscopy (Experimental): Colonoscopy performed with AmplifEYE equipped
  Interventions: Device: AmplifEYE
- Standard colonoscopy (No Intervention): Standard colonoscopy performed

INTERVENTIONS:
Device: AmplifEYE — AmplifEYE colonoscopy
  Arms: AmplifEYE colonoscopy

SUMMARY:
Colonoscopy screening is proven to reduce mortality rates for colorectal cancer, which relies on early detection and removal of colonic polyps. AmplifEYE is a FDA-approved device with a row of flexible detection arms attached to the tip of colonoscope which can separate colonic folds during scope withdrawal and is believed to improve polyp detection. Real-life clinical data on this relatively new device is lacking and this study aims to compare the adenoma and polyp detection rates in AmplifEYE-assisted colonoscopy versus standard colonoscopy.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study. Patients admitted to Queen Elizabeth Hospital and Our Lady of Maryknoll Hospital for colonoscopy are randomly allocated 1:1 to receive either colonoscopy equipped with AmplifEYE (AC) or standard colonoscopy (SC). All study team members will have a prior run-in phase of performing at least 5 AmplifEYE colonoscopies before starting the study. The colonic polyp detection rate (PDR), adenoma detection rate (ADR), serrated polyp detection rate (SDR), caecal intubation time, colonoscope withdrawal time, procedure pain and any adverse events were analyzed in each group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 to 79 years old
* Scheduled for screening, surveillance or diagnostic colonoscopy

Exclusion Criteria:

* Colonic strictures
* History of bowel surgery
* Per-rectal bleeding within six weeks
* Inflammatory bowel disease
* Pregnancy

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 1 day
  number of patients in whom at least one adenoma could be found

SECONDARY OUTCOMES:
Polyp detection rate | 1 day
  number of patients in whom at least one polyp could be found
Serrated polyp detection rate | 1 day
  number of patients in whom at least one serrated polyp could be found
caecal intubation rate | 1 day
  number of patients in whom caecal intubation is acheived
caecal intubation time | 1 day
  time beginning with the insertion of the colonoscope until reaching the caecum

CONTACTS AND LOCATIONS:
Overall Officials: Shun Fung Sze, MBBS, Principal Investigator — Department of Medicine, Queen Elizabeth Hospital
Locations (1):
- Department of Medicine, Queen Elizabeth Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nishihara R, Wu K, Lochhead P, Morikawa T, Liao X, Qian ZR, Inamura K, Kim SA, Kuchiba A, Yamauchi M, Imamura Y, Willett WC, Rosner BA, Fuchs CS, Giovannucci E, Ogino S, Chan AT. Long-term colorectal-cancer incidence and mortality after lower endoscopy. N Engl J Med. 2013 Sep 19;369(12):1095-105. doi: 10.1056/NEJMoa1301969. PMID 24047059
- [Background] Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, Lehman GA, Mark DG. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies. Gastroenterology. 1997 Jan;112(1):24-8. doi: 10.1016/s0016-5085(97)70214-2. PMID 8978338
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133
- [Background] Sawatzki M, Meyenberger C, Marbet UA, Haarer J, Frei R. Prospective Swiss pilot study of Endocuff-assisted colonoscopy in a screening population. Endosc Int Open. 2015 Jun;3(3):E236-9. doi: 10.1055/s-0034-1391418. Epub 2015 Feb 27. PMID 26171436
- [Background] van Doorn SC, van der Vlugt M, Depla A, Wientjes CA, Mallant-Hent RC, Siersema PD, Tytgat K, Tuynman H, Kuiken SD, Houben G, Stokkers P, Moons L, Bossuyt P, Fockens P, Mundt MW, Dekker E. Adenoma detection with Endocuff colonoscopy versus conventional colonoscopy: a multicentre randomised controlled trial. Gut. 2017 Mar;66(3):438-445. doi: 10.1136/gutjnl-2015-310097. Epub 2015 Dec 16. PMID 26674360